CLINICAL TRIAL: NCT06128850
Title: Examining Peri-İmplant and Periodontal Conditions Co-occur: A Cross-Sectional Study
Brief Title: Peri-implant Conditions Mimic Periodontal Conditions
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Other Study IDs: 2022/163
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Peri-implant Health; Periodontitis; Gingivitis
MeSH Terms: conditions — Peri-Implantitis; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peri-implantitis
  Interventions: Other: disease
- Peri-implant mucositis
  Interventions: Other: disease
- Peri-implant health
  Interventions: Other: disease

INTERVENTIONS:
Other: disease — compare to diseases

SUMMARY:
Except for patients with referred clinical bruxism and uncontrolled medical conditions, the study included 123 implants with implanted fixed prostheses that had lasted at least six months after functional prosthetic loading. In all implant patients, the health scale ranged from implants and natural teeth to plaque, gingival index, bleeding in the probe, mouth depth, loss of clinical attachment, and dental implants. The health and illness of the implants have been determined. Patients were divided into three groups: peri-implantitis, peri-implant mucositis, and peri-implant health.

Inclusion Criteria:

* Patients between the ages of 18- 70
* Drugs that have a systemically healthy and controlled treatment situation
* Drivers who have implant-supported fixed prostheses that have been at least six months after functional prosthetic loading Among these groups, it was checked whether periodontitis was seen in patients with peri-implantitis, gingivitis in patients with peri-implant mucositis, and whether healthy gums were seen in individuals with peri-implant health.

To determine the health and disease status of individuals' implants, plaque index (Silness Loe 1964), gingival index (Loe Silness 1963), bleeding on probing (Ainoma Bay 1975), pocket depth measurements, and clinical attachment level were collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18- 70
* Drugs that have a systemically healthy and controlled treatment situation
* Drivers who have implant-supported fixed prostheses that have been at least six months after functional prosthetic loading

Exclusion Criteria:

* Bruxism
* Uncontrolled medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The health and illness of the implants have been determined. Patients were divided into three groups: peri-implantitis, peri-implant mucositis, and peri-implant health.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Plaque index | Baseline
  The plaque index assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth
Gingival index | Baseline
  This measurement is based on the presence or absence of bleeding on gentle probing
Bleeding on probing | Baseline
  Bleeding, leading sign of inflammation inside the connective tissue, is a critical factor for pocket depth measurements, and with other variable factors prevents making reproducible measurements.

SECONDARY OUTCOMES:
Periodontal pocket depth | Baseline
  a pathologically deepened gingival sulcus around a tooth at the gingival margin.
Clinical attachment level | Baseline
  CAL is calculated by subtracting the gingival margin level from the probing depth.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided